CLINICAL TRIAL: NCT06241599
Title: A Multi-center, Randomized, Double-blind, Phase II/III Clinical Trial of AK104 or Placebo in Combination With Chemotherapy as Second-line or More Lines for Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-FXY-023
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AK104 (Experimental): AK104: 6mg/kg intravenous infusion for more than 60 minutes
  Interventions: Drug: GP/PFLL+AK104
- Placebo (Placebo Comparator): placebo: 6mg/kg intravenous infusion for more than 60 minutes
  Interventions: Drug: GP/PFLL+placebo

INTERVENTIONS:
Drug: GP/PFLL+AK104 — Groups 1 and 2: Patients who have not been treated with PFLL in front-line therapy. 5-Fu:200mg/m2/d, d1-30, continuous intravenous infusion; Cisplatin: 80mg/m2, intravenous infusion for 4h, the first and 28th days of each cycle; AK104: 6mg/kg intravenous infusion for more than 60 minutes, used on days 1, 15, 30, 45 of each cycle, and administered 30 minutes before chemotherapy drugs during chemotherapy.
  Groups 3 and 4: Patients who had never used GP in their front-line treatment regimen. Gemcitabine: 1000mg/m2, used on the 1st and 8th day of each cycle; Cisplatin: 80mg/m2 on the first day of each cycle; AK104 6mg/kg intravenous infusion for more than 60 minutes was used on day 1, 15 (single cycle)/or day 8 (double cycle) of each cycle, and was administered 30 minutes before chemotherapy drugs during chemotherapy. Every 3 weeks is a treatment cycle, with a maximum of 6 cycles used. After 6 cycles of chemotherapy, both groups could continue to receive AK104 (once every 2 weeks).
  Arms: AK104
Drug: GP/PFLL+placebo — Groups 1 and 2: Patients who have not been treated with PFLL in front-line therapy. 5-Fu:200mg/m2/d, d1-30, continuous intravenous infusion; Cisplatin: 80mg/m2, intravenous infusion for 4h, the first and 28th days of each cycle; placebo: 6mg/kg intravenous infusion for more than 60 minutes, used on days 1, 15, 30, 45 of each cycle, and administered 30 minutes before chemotherapy drugs during chemotherapy.
  Groups 3 and 4: Patients who had never used GP in their front-line treatment regimen. Gemcitabine: 1000mg/m2, used on the 1st and 8th day of each cycle; Cisplatin: 80mg/m2 on the first day of each cycle; placebo 6mg/kg intravenous infusion for more than 60 minutes was used on day 1, 15 (single cycle)/or day 8 (double cycle) of each cycle, and was administered 30 minutes before chemotherapy drugs during chemotherapy. Every 3 weeks is a treatment cycle, with a maximum of 6 cycles used. After 6 cycles of chemotherapy, both groups could continue to receive placebo (once every 2 weeks).
  Arms: Placebo

SUMMARY:
To compare whether AK104 combined with GP or PFLL can improve survival benefit, safety and tolerability in nasopharyngeal carcinoma patients who have failed first-line treatment; To compare the survival benefits of GP or GFLL treatment in nasopharyngeal carcinoma patients who had failed first-line therapy; To compare the survival benefits of GP or GFLL combined with AK104 in patients with nasopharyngeal carcinoma who had failed first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years; 2. Non-keratinized differentiated or undifferentiated nasopharyngeal carcinoma confirmed by pathology; 3. For patients with recurrent and metastatic nasopharyngeal carcinoma who are not eligible for local treatment and meet the definition of the staging system (8th edition) of the International Union against Cancer and the American Joint Committee on Cancer (UICC/AJCC), local treatment mainly refers to measures related to anti-tumor treatment, including surgery, radiofrequency ablation, transhepatic arterial chemoembolization (TACE), radiotherapy (except for patients with bone metastasis). A locally appropriate dose of radiotherapeutic therapy for symptomatic relief) 4. Patients with nasopharyngeal carcinoma recurrence and metastasis who failed first-line treatment; 5.ECOG performance score 0 or 1; 6. There is at least one measurable lesion according to the RECIST1.1 evaluation criteria, and a lesion that has previously received, for example, radiation therapy can be considered a target lesion if there is objective evidence of disease progression. 7. Patients are required to provide tissue samples within three years prior to enrollment; 8. Expected survival ≥3 months; 9. The functions of vital organs meet the following requirements (no blood components, cell growth factors, whitening drugs, thrombocytophytics, or anemia correction drugs are allowed within 14 days before screening) : · Neutrophil absolute count (ANC) ≥1.5×109/L· Platelets ≥100×109/L; · Hemoglobin ≥8.0g/dl (note: Hemoglobin ≥8.0g/dl through blood transfusion or other intervention is acceptable); · Serum albumin ≥2.8g/dL; · Bilirubin ≤ 1.5x ULN, ALT and AST≤ 1.5x ULN; If there is liver metastasis, ALT and AST are less than 5 times ULN. Creatinine clearance ≥50mL/min (using the standard CockcroftGault formula, see Annex II); 10. Women of reproductive age who have an unsterilized sexual partner should use at least one highly effective form of birth control; 11. Unsterilized men with a partner of childbearing age must use a highly effective form of birth control from day 1 to day 120 of the last use of the study drug; 12. Informed consent has been signed.

Exclusion Criteria:

1. Previous history of allergy to 5-Fu, cisplatin, gemcitabine, other monoclonal antibodies or any component of CTLA-4 and PD1 bispecial antibodies; In the past, CTLA-4 and PD1-specific antibody therapy were used simultaneously. 2. Had major surgery other than diagnosis of nasopharyngeal cancer within 28 days prior to randomization or was expected to require major surgery during the study period; 3. The subject has any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or asthma that has been in complete remission in childhood can be adults without any intervention.Patients with asthma requiring medical intervention with bronchodilators were not included); 4. Subjects were taking immunosuppressants, or systemic, or absorbable local hormone therapy for immunosuppressive purposes (doses >10mg/ day of prednisone or other therapeutic hormones) and continued to use within 2 weeks prior to enrollment; 5. Known subject is previously allergic to macromolecular protein preparation ingredients; 6. The subject has clinically symptomatic central nervous system metastases (e.g. brain edema, need for hormonal intervention, or progression of brain metastases); Other aggressive malignancies within 7.5 years, except locally curable (appearing to cure) malignancies such as basal or squamous cell carcinoma of the skin, superficial cancers of the bladder, cervix and breast in situ; 8. Active autoimmune disease requiring systemic treatment within the last two years, except vitiligo, alopecia, Grave disease, psoriasis or eczema that did not require systemic treatment within the last two years, hypothyroidism requiring stable hormone replacement therapy only (due to autoimmune thyroiditis), type 1 diabetes requiring stable dose insulin replacement therapy only; Childhood asthma that has been completely cured in adulthood without intervention or primary disease that does not recur unless stimulated by external factors; 9. Active or previous inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea); 10. Systemic glucocorticoid therapy (dose equivalent to 10mg/ day of prednisone) or other immunosuppressants are required within the first seven days of initial administration of the investigational drug. 11. Having allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 12. Gastrointestinal perforation or fistula within the first six months of enrollment; 13. There were necrotic foci within the first four weeks of enrollment that researchers thought might be a potential source of major bleeding;14. History of interstitial pneumonia; 15. History of active tuberculosis; 16. Serious infections, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia, occur within four weeks prior to the first application of the investigational drug; 17. Active infections that require systematic treatment; 18. Untreated chronic hepatitis B or chronic HBVDNA≥1000IU/ml or active hepatitis C. Non-active HBsAg carriers, stable hepatitis B after treatment (HBVDNA < 1000IU/ml) and cured hepatitis C can be included. Patients who are positive for HCV antibodies can only be enrolled if they test negative for HCVRNA. 19. History of major surgery within 30 days before the first application of the investigational drug; 20. There is meningeal metastasis or active brain metastasis; 21. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage; 22. Toxicity problems unresolved at the time of previous antitumor therapy, defined as unresolved to level 0 or 1 of NCICTCAEv5.0, or levels specified in the inclusion/exclusion criteria, except hair loss. 23. Live attenuated vaccines were administered within 30 days prior to the first application of the investigational drug, or live attenuated vaccines were planned to be administered during the study period. 24. Known history of severe allergy to other monoclonal antibodies; 25. Pregnant or lactating women; 26. Have clinical symptoms or diseases of heart that are not well controlled, such as: ① heart failure of NYHA2 or above; ② Unstable angina pectoris; ③ Myocardial infarction occurred within 1 year; Patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; 27. Subjects had an active infection or unexplained fever >38.5 degrees during screening or prior to initial dosing (as determined by the investigator, subjectsFever due to tumor can be included in the group); •28. Allergic to AK104 ingredients; 29. The subject has a known history of psychotropic substance abuse, alcohol abuse, or drug use; 30. According to the investigator's judgment, the subjects have other factors that may lead to the forced termination of the study, such as other serious illnesses (including mental illness) requiring combined treatment, serious abnormalities in laboratory tests, and family or social factors that may affect the safety of the subjects, or the collection of test data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  Progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes